CLINICAL TRIAL: NCT06096493
Title: Predictors of Disease Free Survival After Curative Cancer Rectum Surgery
Brief Title: Prognostic Factors Affecting Recurrence and Disease-Free Survival After Surgical Resection for Cancer Rectum
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Abdallah Mohamed Taha Aly, Assistant Professor of general Surgery, South Valley University
Other Study IDs: SVU-MED-SUR011-4-23-4-621
Record Dates: First submitted 2023-10-19; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Rectal Cancer
Keywords: cancer rectum; recurrence; disease free survival
MeSH Terms: conditions — Rectal Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cancer rectum underwent curative surgery: Patients with cancer rectum underwent curative surgery
  Interventions: Procedure: curative surgery for cancer rectum

INTERVENTIONS:
Procedure: curative surgery for cancer rectum — Curative surgery for cancer rectum.

SUMMARY:
Tumor recurrence after curative surgical resection for rectal cancer is a serious complication that greatly affects the overall morbidity and the outcome. This study aims to identify the different prognostic factors affecting recurrence and disease-free survival after surgery.

DETAILED DESCRIPTION:
A retrospective analysis of patients operated for cancer rectum with curative intent from.

Exclusion criteria will include patients with familial adenomatous polyposis, multiple synchronous or metachronous rectal cancers, and death within 3 months. Incomplete patients' files and patients that lost follow-up will be excluded.

Demographic, histopathological, follow up and outcome data will be collected from completed patients' files. Demographics include age, gender, family history, and chief complaint at the presentation. Histopathological data include tumor grade, vascular-perineural invasion, the total number of lymph nodes removed, and positive lymph nodes.

Lymph node ratio will be defined as the ratio of positive lymph nodes to the total number of retrieved lymph nodes in a histopathology specimen. Disease-free survival will be calculated for each patient based on the time of surgery to the time of recurrence detection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had curative surgery for cancer rectum.

Exclusion Criteria:

* Patients with familial adenomatous polyposis (FAP), multiple synchronous or metachronous rectal cancers, and death within 3 months
* Patients that lost follow-up will be excluded.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - Patients who had curative surgery for cancer rectum.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Tumor recurrence | Through study completion, an average of 3 year
  Presence of Tumor recurrence after curative surgery for cancer rectum.
Disease free survival. | up to 5 years
  From date of surgery until the date of recurrence detection.

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah M Taha, MD, Principal Investigator — South Valley University, Egypt.
Locations (1):
- Qena Faculty of Medicine, South Valley University Hospitals, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He WZ, Xie QK, Hu WM, Kong PF, Yang L, Yang YZ, Jiang C, Yin CX, Qiu HJ, Zhang HZ, Zhang B, Xia LP. An increased number of negative lymph nodes is associated with a higher immune response and longer survival in colon cancer patients. Cancer Manag Res. 2018 Jun 18;10:1597-1604. doi: 10.2147/CMAR.S160100. eCollection 2018. PMID 29950897
- [Background] Li Destri G, Di Carlo I, Scilletta R, Scilletta B, Puleo S. Colorectal cancer and lymph nodes: the obsession with the number 12. World J Gastroenterol. 2014 Feb 28;20(8):1951-60. doi: 10.3748/wjg.v20.i8.1951. PMID 24587671
- [Background] Hashiguchi Y, Muro K, Saito Y, Ito Y, Ajioka Y, Hamaguchi T, Hasegawa K, Hotta K, Ishida H, Ishiguro M, Ishihara S, Kanemitsu Y, Kinugasa Y, Murofushi K, Nakajima TE, Oka S, Tanaka T, Taniguchi H, Tsuji A, Uehara K, Ueno H, Yamanaka T, Yamazaki K, Yoshida M, Yoshino T, Itabashi M, Sakamaki K, Sano K, Shimada Y, Tanaka S, Uetake H, Yamaguchi S, Yamaguchi N, Kobayashi H, Matsuda K, Kotake K, Sugihara K; Japanese Society for Cancer of the Colon and Rectum. Japanese Society for Cancer of the Colon and Rectum (JSCCR) guidelines 2019 for the treatment of colorectal cancer. Int J Clin Oncol. 2020 Jan;25(1):1-42. doi: 10.1007/s10147-019-01485-z. Epub 2019 Jun 15. PMID 31203527
- [Background] Heald RJ, Husband EM, Ryall RD. The mesorectum in rectal cancer surgery--the clue to pelvic recurrence? Br J Surg. 1982 Oct;69(10):613-6. doi: 10.1002/bjs.1800691019. PMID 6751457
- [Background] Tschmelitsch J, Kronberger P, Glaser K, Klingler A, Bodner E. Survival after surgical treatment of recurrent carcinoma of the rectum. J Am Coll Surg. 1994 Jul;179(1):54-8. PMID 8019725
- [Background] Feeney G, Sehgal R, Sheehan M, Hogan A, Regan M, Joyce M, Kerin M. Neoadjuvant radiotherapy for rectal cancer management. World J Gastroenterol. 2019 Sep 7;25(33):4850-4869. doi: 10.3748/wjg.v25.i33.4850. PMID 31543678